CLINICAL TRIAL: NCT06156475
Title: The Effect of Electromyographic Biofeedback and Proprioception Exercises on Pain and Functionality in Patients With Subacromial Impingement Syndrome: A Randomized Controlled Study
Brief Title: The Physiotherapy Approaches in Patients With Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Kaya Mutlu, PT, Prof. Dr., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Istanbul Aydin University
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-11

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Shoulder impingement syndrome; shoulder pain; proprioception; biofeedback
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: The study consisted of patients with subacromial impingement syndrome evaluated by an orthopedist. Patients who met the inclusion criteria were divided into two groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioception Exercise Group (Experimental): Wand exercises and Proprioception exercises
  Interventions: Procedure: Proprioception exercises; Procedure: Wand Exercise
- Proprioception exercises with Electromyographic Biofeedback (Active Comparator): Wand exercises and Proprioception exercises with Electromyographic Biofeedback
  Interventions: Procedure: Proprioception exercises with Electromyographic Biofeedback; Procedure: Wand Exercise

INTERVENTIONS:
Procedure: Proprioception exercises — Patients trained for proprioception exercises.
  Arms: Proprioception Exercise Group
Procedure: Proprioception exercises with Electromyographic Biofeedback — Patients trained for Proprioception exercises with Electromyographic Biofeedback
  Arms: Proprioception exercises with Electromyographic Biofeedback
Procedure: Wand Exercise — Patients were educated with wand exercises.

SUMMARY:
The aim of this study is to investigate the effectiveness of Electromyographic Biofeedback with proprioception exercises on pain, range of motion, muscle strength, proprioception and functionality in patients with subacromial impingement syndrome.

DETAILED DESCRIPTION:
This study is planned as a prospective, randomized clinical study. Patients with subacromial impingement syndrome who volunteered to participate in the study, met the inclusion criteria, and signed the consent form were randomly assigned to the proprioception exercise group and the proprioception exercise with electromyographic biofeedback group. Demographic and clinical data of the patients were recorded. Shoulder function with Disabilities of the Arm, Shoulder and Hand scale, pain with VAS, painless active shoulder flexion, abduction, and external-internal rotation with goniometer, muscle strength with Manual Muscle Tester, proprioception (55°-90°- 125° angles of flexion and abduction, and angular deviations) with the Laser-pointer assisted angle reproduction test were evaluated, and patient satisfaction was evaluated with The Global Rating of Change Scale. After the initial evaluations were completed, only proprioception exercises and proprioception exercises with EMG-BF were applied 2 days a week for 8 weeks. Additionally, both groups were given Want exercises.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with subacromial impingement syndrome,
* Being between the ages of 18 and 65,
* Not having received medical treatment,
* Not having received a shoulder-related physiotherapy program in the last year,
* Not having had any shoulder-related surgery,

Exclusion Criteria:

* Neurological deficits of the upper extremity and the presence of another orthopedic disorder, rheumatic or congenital disease other than subacromial impingement syndrome,
* Presence of mental problem,
* Having received corticosteroid treatment in the last year,
* Upper extremity fracture,
* Acute cervical pathology,
* Having cardiovascular and systemic diseases that prevent working,
* Pregnancy,
* Those with communication problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand scale | 8 weeks
  The Disabilities of the Arm, Shoulder and Hand scale was used to measure shoulder function. The Disabilities of the Arm, Shoulder and Hand scale consists of 30 items. The total score that can be obtained from items scored between 1-5 varies between 0-100. An increase in the score indicates a decrease in function.

SECONDARY OUTCOMES:
Visual analogue scale | 8 weeks
  The severity of pain was measured Visual analogue scale. ccording to this scale, patients rated their pain between 0 and 10. As the score increases, the pain increases.
Joint range of motion | 8 weeks
  Active shoulder flexion, abduction, and external-internal rotation range of motion was measured with goniometer.
Muscle strength | 8 weeks
  Shoulder flexion, abduction, and external-internal rotator muscle strength was measured with manual muscle tester.
Proprioception | 8 weeks
  To evaluate joint position sense, laser pointer-assisted angle reproduction test was applied for measurements at 55°-90°-125° flexion and abduction angles.
Patient satisfaction | 8 weeks
  The amount of improvement or deterioration in patients was assessed with the "Global Rating Change Scale".This scale is scored according to a 7-point Likert type (-3: much worse, -2: worse, -1: slightly worse, 0: the same, 1: slightly better, 2: quite better, 3: much better).

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Kaya Mutlu, Professor, Principal Investigator — Bandırma Onyedi Eylül University; Buse Aydin, M.Sc., Study Chair — Istabul Aydin University; Yasemin Karaaslan, Asst. Prof., Study Chair — Mustafa Kemal University; Hanifegül Taskiran, Professor, Study Chair — Istanbul Aydın University; Nezih Ziroglu, MD, Study Chair — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Istanbul Aydin University, Istanbul, Florya, Turkey (Türkiye)